CLINICAL TRIAL: NCT06318819
Title: Plaque Removal Effectiveness of a Flossing Device (Dental Floss Holders) Compared to the Conventional Flossing in Adults: a Randomized Clinical Trial.
Brief Title: Plaque Removal Effectiveness of a Flossing Device Compared to the Conventional Flossing in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maha A. Bahammam (Other)
Collaborators: King Abdulaziz University (Other)
Responsible Party: Sponsor-Investigator, Maha A. Bahammam, Professor, King Abdulaziz University
Organization: King Abdulaziz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 159-11-19.
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Tooth Decay; Cavities of Teeth; Gingivitis; Plaque
Keywords: Plaque Removal; Flossing Device
MeSH Terms: conditions — Dental Caries; Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental Floss Holders (Experimental): Dental Floss Holders was constructed.
  Interventions: Device: Dental Floss Holders
- conventional flossing (Active Comparator): conventional flossing to the opposite arch.
  Interventions: Device: Dental Floss Holders

INTERVENTIONS:
Device: Dental Floss Holders — Dental Floss Holders for flossing purposes

SUMMARY:
* Objective: To evaluate the effectiveness in plaque removal of the new device; Dental floss holders and compare the results to the conventional way of flossing.
* Methods: Thirty adult male and female participants participated in this randomized, single-use, single-blind clinical study. Participants were randomly assigned to one of two groups; Group A: Consists of 30 participants in whom Dental Floss Holders (DFH) was constructed to either maxillary or mandibular arch randomly. Group B: Consists of 30 participants in whom conventional flossing (CF) was done to the other arch.

Participants attended the first visit for primary impression taking in order to construct the DFH. In the second visit, participants were examined by a blinded examiner to record their plaque index using O'Leary index. Then, they flossed using DFH and CF according to the group they were assigned to. Participants were monitored to ensure proper coverage of all the areas following precise instructions. They then brushed their teeth for approximately 2 minutes using modified bass technique. Next, plaque index was recorded again using the O'leary index. Time was recorded during flossing of each arch. Finally, participants were given a questionnaire to assess their satisfaction of the device.

* Results: The differences between the groups showed the DFH group with a 62.8% reduction in whole mouth plaque and 63.3% for proximal plaque compared to 52.9% and 50.4% for the CF group, respectively (p = 0.01). The DFH was more time efficient in removing plaque from the marginal regions with an average time of 00:00:37 in comparison to the CF which averaged in 00:02:07 (p < 0.001). A total of 26 participants (86.7%) preferred using the DFH over the CF.
* Conclusion: With the combination of toothbrushing, the Dental Floss Holders is significantly more effective and time efficient than conventional flossing in removing plaque from tooth surfaces.

ELIGIBILITY:
1. Able to understand, read, and write in Arabic or English and provide written informed consent prior to participation.
2. Not engaged in any other clinical study during the day of examination.
3. Non-smoker and in good general health.
4. Does not have any systemic disease that influences the oral tissue (e.g., diabetes, autoimmune disease, medication/antibiotics).
5. Fully dentate (not including 3rd molars) with established proximal contacts.
6. Good oral health with no hard or soft tissue lesions, no gross caries, no probing depths greater than 4 mm, no obvious advanced periodontal disease, no fixed orthodontic appliances, nor removable partial dentures.
7. Does not have any dexterity limitation.
8. Not pregnant at the time of the study.

Ages: 20 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Dental Floss Holders (DFH) | 6 months
  62.8% reduction in whole mouth plaque 63.3% for proximal plaque
Conventional flossing (CF) | 6 months
  52.9% reduction in whole mouth plaque and 50.4% for proximal plaque

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Thirty adult male and female participants participated in this randomized, single-use, single-blind clinical study. Participants were randomly assigned to one of two groups; Group A: Consists of 30 participants in whom Dental Floss Holders (DFH) was constructed to either maxillary or mandibular arch randomly. Group B: Consists of 30 participants in whom conventional flossing (CF) was done to the other arch.
  Participants attended the first visit for primary impression taking in order to construct the DFH. In the second visit, participants were examined by a blinded examiner to record their plaque index using O'Leary index. Then, they flossed using DFH and CF according to the group they were assigned to. Next, plaque index was recorded again using the O'leary index. Time was recorded during flossing of each arch.